CLINICAL TRIAL: NCT03662568
Title: A Open-label, Single Center Drug Interaction Study of Morphothiadine Mesilate/Ritonavir , Entecavir and Tenofovir Disoproxil Fumarate in Healthy Subjects
Brief Title: A Drug-drug Interaction (DDI) Study of Morphothiadine Mesilate/Ritonavir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DGLS4-18-001
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2018-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A:Group A (Experimental): Subjects will receive GLS4+RTV on Day 1,followed by ETV on Day11-21 and co-administration with GLS4+RTV on Day 21.
  Interventions: Drug: GLS4; Drug: RTV; Drug: ETV
- Part A:Group B (Experimental): Subjects will receive ETV on Day 1,followed by GLS4+RTV on Day11-21 and co-administration with ETV on Day 21.
  Interventions: Drug: GLS4; Drug: RTV; Drug: ETV
- Part B:Group C (Experimental): Subjects will receive GLS4+RTV on Day 1,followed by TDF on Day11-21 and co-administration with GLS4+RTV on Day 21.
  Interventions: Drug: GLS4; Drug: RTV; Drug: TDF
- Part B:Group D (Experimental): Subjects will receive TDF on Day 1,followed by GLS4+RTV on Day11-21 and co-administration with TDF on Day 21.
  Interventions: Drug: GLS4; Drug: RTV; Drug: TDF

INTERVENTIONS:
Drug: GLS4 — Administered GLS4 120 mg orally three times daily in fed state
  Other Names: Morphothiadine Mesilate Capsules
Drug: RTV — Administered RTV 100 mg orally three times daily in fed state
  Other Names: Ritonavir tablet
Drug: ETV — Administered orally ETV 0.5 mg once daily in fasted state
  Other Names: Entecavir table
  Arms: Part A:Group A; Part A:Group B
Drug: TDF — Administered TDF 300 mg orally once daily in fasted state
  Other Names: Tenofovir Disoproxil Fumarate table
  Arms: Part B:Group C; Part B:Group D

SUMMARY:
The purpose of this study is to evaluate the drug-drug-interaction (DDI), pharmacokinetics (PK) and tolerability of Morphothiadine Mesilate/Ritonavir combined with Entecavir or Tenofovir Disoproxil Fumarate in healthy subjects

DETAILED DESCRIPTION:
This is a 2-part study with each part is an open-label, crossover study in healthy adult subjects.

Total 56 subjects will be enrolled into the study and divided into 2 part (Part A and Part B), 28 subjects in each part. Part A is to evaluate the drug-interaction between GLS4/RTV and ETV, Part B is to evaluate the drug-interaction between GLS4/RTV and TDF. With each part, the subject will be split into two groups and receive study drug per the defined treatment periods of Day 1, Day 11-20 and Day 21.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions
* Be able to complete the study according to the trail protocol
* Subjects (including partners) have no pregnancy plan within 1 year after the last dose of study drug and voluntarily take effective contraceptive measures
* Male subjects and must be 18 to 45 years of age inclusive
* Body weight ≥ 50 kg and body mass index（BMI）between 18 and 28 kg / m2, inclusive
* Physical examination and vital signs without clinically significant abnormalities.

Exclusion Criteria:

* Use of >5 cigarettes per day during the past 3 months
* Known history of allergy to study drugs，or allergies constitution ( multiple drug and food allergies)
* History of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits or 100 mL of wine)
* Donation or loss of blood over 450 mL within 3 months prior to screening
* 12-lead ECG with clinically significant
* Positive for Viral hepatitis (including hepatitis B and C), HIV and syphilis
* Subjects deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1-2 and Day 21-23
  Maximum plasma concentration of study drugs
AUC | Day 1-2 and Day 21-23
  Area under the plasma concentration-time curve of study drugs
Tmax | Day 1-2 and Day 21-23
  Time to maximum concentration of study drugs
T1/2 | Day 1-2 and Day 21-23
  Terminal half-life of study drugs
Adverse events | Baseline to day 23
  To assess the safety and tolerability after dosing

SECONDARY OUTCOMES:
CL/F | Day 1-2 and Day 21-23
  Apparent clearance of study drugs
Vz/F | Day 1-2 and Day 21-23
  Apparent volume of distribution of study drugs
Cmin | Day 1-2 and Day 21-23
  Minimum plasma concentration of study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China